CLINICAL TRIAL: NCT04574830
Title: Clinical Survey Study to Evaluate Biomarkers and Clinical Manifestations in Individuals With Glycogen Storage Disease Type III (GSD III)
Brief Title: Study to Evaluate Biomarkers and Clinical Manifestations in Individuals With Glycogen Storage Disease Type III (GSD III)
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX053-CL001
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Glycogen Storage Disease Type III
MeSH Terms: conditions — Glycogen Storage Disease Type III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The primary objective of this study is to evaluate potential biomarkers of GSD III.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed historical diagnosis of GSD III based on pathogenic mutations in the AGL gene on both alleles or GDE deficiency based on biopsy of liver, muscle, or fibroblasts
* Willing to comply with all study procedures
* Willing and able to provide written informed consent. If a minor, willing and able to provide written assent and have a legally authorized representative willing and able to provide written informed consent

Exclusion Criteria:

* Presence or history of any condition that, in the view of the Investigator, places the subject at high risk of poor study compliance, interferes with study participation, or interferes with the subject's ability to safely or reliably complete the study assessments
* Use of any IP within 30 days prior to informed consent/assent or at the time of enrollment

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a confirmed diagnosis of GSD III
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Urine hexose tetrasaccharide (Hex4): mean and variance | Up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (4):
- United States (4):
  - University of California, Irvine, California
  - Children's Hospital Orange County, Orange, California
  - Colorado Children's Hospital, Aurora, Colorado
  - University of Texas Medical School, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy/GSD III Disease Information — https://ultrarareadvocacy.com/glycogen-storage-disease-type-iii-gsdiii/